CLINICAL TRIAL: NCT05159115
Title: Sucrase-isomaltase Deficiency as a Cause of Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED 358
Record Dates: First submitted 2021-12-06; First posted 2021-12-15 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-11

CONDITIONS: Irritable Bowel Syndrome; Sucrose Intolerance Due to Sucrase-Isomaltase Deficiency; Carbohydrate; Malabsorption; Sucrase Isomaltase Deficiency; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Malabsorption Syndromes; Sucrase-isomaltase deficiency, congenital; Gastrointestinal Diseases | interventions — FODMAP Diet; Starch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-FODMAP diet (Active Comparator): Patients with IBS on a 4-week low-FODMAP diet.
  Interventions: Other: Low-FODMAP diet
- Starch- and Sucrose Reduced Diet (Experimental): Patients with IBS on a s 4-week Starch- and Sucrose Reduced Diet (SSRD).
  Interventions: Other: Starch- and Sucrose Reduced Diet (SSRD)

INTERVENTIONS:
Other: Low-FODMAP diet — 4 weeks of a diet low in fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAPs)
  Arms: Low-FODMAP diet
Other: Starch- and Sucrose Reduced Diet (SSRD) — 4 weeks of a diet low in starch and sucrose
  Arms: Starch- and Sucrose Reduced Diet

SUMMARY:
Irritable bowel syndrome (IBS) is a functional disorder causing troublesome symptoms and reduced quality of life. It affects 10-20% of the population, hence creates large costs for society. About 30-40% of all IBS patients do not benefit from current treatment options. Sucrase-isomaltase (SI) deficiency is an unexplored condition, that may explain symptoms in IBS patients who experience no effect from today's treatments. Currently, a duodenal biopsy is the gold standard for the diagnosis of SI deficiency, however the condition is not well investigated. A 13C-labelled breath test holds promise as a non-invasive alternative, but it has not previously been validated.

This project will address the knowledge gap related to a possible association between SI deficiency and IBS by addressing two research questions that have never been answered before. We aim to:

1. Validate the 13C-labelled breath test as a diagnostic tool by assessing the strength of the association between the breath test and SI activity measured in duodenal biopsies
2. Use the 13C-labelled breath test in a randomized dietary crossover trial comparing a starch and sucrose reduced diet (SSRD) with the standard low-FODMAP diet in IBS patients, to evaluate whether SI activity is associated with dietary changes according to symptom severity and gut microbiota composition

DETAILED DESCRIPTION:
The projects includes two studies:

Study 1: Validation of the 13C-labelled breath test to diagnose sucrase-isomaltase deficiency

Background: In order to validate the 13C-sucrose breath test to diagnose SI deficiency, the test result must be compared to the "gold standard" method for diagnosis; i.e. measurements of enzyme activity from intestinal biopsies by "The Dahlquist Method", and a reference material must be established.

Objective: To compare results from the 13C-labelled breath test to enzyme activity measured in biopsies collected from the proximal small intestine in a limited patient group referred for a gastroscopic examination.

Design: A cross-sectional study.

Primary endpoint: SI activity as measured with a breath test and enzyme activity with assay of biopsy material.

Recruitment and patient characteristics: Patients referred for gastroscopic examination with duodenal biopsies and with suspected GI disorder, will be included consecutively.

Sample size: We aim to include 40 patients. No studies validating breath test results in our patient group are available. However, based on preliminary results suggesting that 35% of IBS patients have SI deficiency,13 we are 95% likely to find between 8 and 21 patients with SI deficiency when examining 40 patients. Assuming 80% concordance between the two methods to (correct proportion of successes), we would need 12 positive cases. Thus, if 40 individuals are included, the study is sufficiently powered (alpha=5% and beta=20%, using McNemar's test of concordance).

Study 2: Sucrase-isomaltase deficiency as a cause of symptoms in patients with irritable bowel syndrome

Objectives: To examine the effect of a 4-week SSRD on GI- and extraintestinal symptoms, gut microbiota composition and fecal fermentation in patients with IBS (with and without SI deficiency), and compare the SSRD with a 4-week low-FODMAP diet to investigate whether the patients with a breath test result indicating SI deficiency respond better to the SSRD than the patients with normal SI activity. Gut microbiota have been suggested to have a central role in IBS etiology, hence evaluation of gut microbiota composition and fecal fermentation will be included to increase the knowledge regarding the effects of dietary change on gut microbiota composition and activity related to SI deficiency.

Design: A randomized, open clinical crossover trial with a dietary intervention in a group of IBS patients, lasting for 4+4 weeks (SSRD vs. low-FODMAP) with a 1-week wash-out period in between. Breath tests will be taken at inclusion, but the results will be "blinded", e.g. not available for anyone conducting the trial before end of the study. A SSRD will be compared to the low-FODMAP diet. All participants will be given dietary advice from a registered clinical dietitian. Briefly, all forms of sucrose-containing foods (e.g. sweets, jam, and cakes) should be avoided, and foods rich in starch should be reduced on the SSRD.

Primary endpoint: Symptom severity by IBS-Symptom Severity Scale (IBS-SSS).

Secondary endpoints: Gut microbiota composition, fecal fermentation measured by short chain fatty acids (SCFAs) and assessment of quality of life by the Patient Reported Outcome Measurement Information System (PROMIS-29).

Recruitment and patient characteristics: IBS patients referred to the outpatient clinic at the Department of Gastroenterology at Lovisenberg Diaconal Hospital for dietary guidance by a registered dietitian will be consecutively included.

Sample size: The primary end point is change in IBS symptom severity (IBS-SSS) at the end of the treatment period relative to baseline, and the proportion of responders to the dietary intervention is based on the recommended cut-off of a reduction (ie, improvement) in total IBS-SSS score of 50 points, which is considered to be clinically meaningful improvement. To plan our sample size, we performed a power calculation based on the ability to detect a difference between the two diets in reduction of IBS-SSS score of at least 50 points with 80% power, assuming an SD of 100. The calculation indicated that we would need 64 patients. To allow for 15-20% drop-out, we aim to include 80 patients.

ELIGIBILITY:
Validation of the 13C-labelled breath test to diagnose sucrase-isomaltase deficiency (n=40)

Inclusion Criteria:

* Signed informed consent
* BMI 18-30 kg/m2
* Referred for gastroscopic examination with suspected GI disorder

Exclusion Criteria:

• Unwilling or not capable of signing the informed consent

Sucrase-isomaltase deficiency as a cause of symptoms in patients with irritable bowel syndrome (n=80)

Inclusion Criteria:

* Signed informed consent
* BMI 18-30 kg/m2
* IBS diagnosis according to Rome IV criteria

Exclusion Criteria:

* Inflammatory bowel disease, celiac disease or diabetes mellitus
* Chronic immune diseases affecting the GI-system
* Unwilling/unable to maintain a stable diet throughout the study period
* Use of antibiotic treatment for the last 4 weeks
* Currently on a restrictive diet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-14 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
IBS symptom severity | 4 weeks
  Symptom severity measured by the IBS-Symptom Severity Scale (IBS-SSS)

SECONDARY OUTCOMES:
Gut microbiota composition | 4 weeks
  Analysis of fecal samples for evaluation of microbiota composition in fecal samples collected at baseline and after each 4-week diet intervention
Fecal fermentation measured by short chain fatty acids (SCFAs) | 4 weeks
  Analysis of SCFAs in fecal samples collected at baseline and after each 4-week diet intervention
Quality of life in IBS | 4 weeks
  Assessment of quality of life by the Patient Reported Outcome Measurement Information System (PROMIS-29)

IPD SHARING:
Plan to Share IPD: No